CLINICAL TRIAL: NCT03765593
Title: Gene Expression of Interferon (INF) and B Lymphocyte Biomarkers as Markers of Systemic Affectation and Lymphoproliferative Disease in Primary Sjögren's Syndrome
Brief Title: Biomarkers in Primary Sjögren's Syndrome
Acronym: pSS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Council of Scientific and Technical Research, Argentina (Other Government)
Responsible Party: Principal Investigator, Maria Soledad Retamozo, Research Assistant, National Council of Scientific and Technical Research, Argentina
Other Study IDs: 3398
Record Dates: First submitted 2018-11-20; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Primary Sjögren Syndrome; Lymphoma, Non-Hodgkin
Keywords: Primary Sjogren Syndrome; Lymphoma; Biomarker
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Salivary gland, saliva, blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Study group 1: Immunopositive primary SS (Anti-SSA +/anti-Ro+) will receive salivary gland biopsy.
  Interventions: Procedure: Biopsy Salivary Gland
- Study group 2: Immunonegative primary SS (Anti-SSA -/anti Ro-, biopsy Chisholm-Mason 3-4) will receive salivary gland biopsy.
  Interventions: Procedure: Biopsy Salivary Gland
- Study group 3: Non-autoimmune sicca syndrome (Anti-SSA/anti Ro-, biopsy Chisholm-Mason 2 o less) will receive salivary gland biopsy.
  Interventions: Procedure: Biopsy Salivary Gland
- Control group: Patients who have sicca syndrome but do not meet the classification criteria of Sjögren's syndrome, therefore, at the time of evaluating these patients to determine whether or not they have the disease are what will serve as controls since according to the usual diagnostic process, the same studies will be carried out as for patients with the proposed disease. Will receive salivary gland biopsy.
  Interventions: Procedure: Biopsy Salivary Gland

INTERVENTIONS:
Procedure: Biopsy Salivary Gland — A minor salivary gland biopsy will be performed at lower lip, with the minimally invasive technique that is carried out in Rheumatology Unit as a routine procedure for the diagnosis of pSS, from there it will be taken between 2-3 glands for the study. RNAlater®(Ambion, Inc., Texas, United States of America) will be stored in solution for the stabilization and preservation of RNA at -80ºC.

SUMMARY:
The clinical spectrum of primary Sjogren Syndrome (pSS)ranges from sicca syndrome to systemic involvement (extraglandular manifestations), including a large number of manifestations that may be the form of presentation or appear after the disease is diagnosed, and that clearly mark the prognosis of the disease.

Gene expression levels of Interferon (INF) and B Lymphocyte Biomarkers as Markers of Systemic Affectation and Lymphoproliferative Disease in, together with clinical and laboratory parameters, will provide significant information about the risk of developing hematological neoplasms in patients with pSS at different stages of the disease, and lead to better management of the disease treatment and therapeutic behaviors.

Using the proposed technique allows us to study the gene expression at the mRNA level of each biomarker, which allows us to anticipate the irreversible changes that take place due to the progress of the pathology in progress, since the molecular changes precede the histological changes and in the pathological diagnosis.

DETAILED DESCRIPTION:
This project, address the value of these proposed biomarkers in pSS with regard to disease activity and risk stratification of pSS subsets. The investigator's group aim to determine if the proposed biomarkers and their gene expression in saliva, peripheral blood and minor salivary gland samples in patients with pSS are increased to know the degree of their usefulness in daily clinical practice, to indicate which patients have a highest risk of developing a hematological malignancy and to know if these biomarkers are useful to recognize patients who have greater activity of the disease to be able to use it in the follow-up of the disease and as a future responder of the new biological therapies against B cells, INF and monocytes.

Gene expression is a highly regulated mechanism that controls the function and adaptability of all living cells. The field of gene expression analysis has undergone important advances in biomedical research. Today, quantification techniques of mRNA expression have led to improvements in the identification of the gene and the sub-classification of the disease, for example, the expression of specific genes (mRNA) can be quantified by reverse transcription and PCR in quantitative real time. This is the most sensitive technique available to detect and quantify mRNA, where extremely small sample sizes can be used in mRNA quantification. Molecular changes precede histological changes and clinicians in the diagnosis of a pathology. For this reason, studying gene expression at the mRNA level allows us to anticipate irreversible changes that take place due to the progress of the pathology in progress.

ELIGIBILITY:
Inclusion Criteria:

* Patients: cross sectionally patients will be included for clinical suspicion of primary SS or with the diagnosis already established in Rheumatology unit.

The following inclusion criteria will be applied to the study:

* Age > 18 years
* Informed consent of the patient.

Exclusion Criteria:

* Impossibility of obtaining consent (cognitive impairment, other causes).
* Associated systemic autoimmune or rheumatological diseases.
* Chronic viral infections (HCV, HBV, HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with sicca and primary Sjogren Syndrome will be recruited from multiple sites.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Gene expression levels in immune cells in salivary gland biopsy samples from participants with and without pSS | Up to 24 months
  To identify a biomarker of disease activity, measured by the real-time PCR reactions (qRT-PCR).
Gene expression levels in immune cells in blood samples from participants with and without pSS | Up to 24 months
  To identify a biomarker of disease activity, measured by the real-time PCR reactions (qRT-PCR).
Gene expression levels in immune cells in saliva samples from participants with and without pSS | Up to 24 months
  To identify a biomarker of disease activity, measured by the real-time PCR reactions (qRT-PCR).

SECONDARY OUTCOMES:
Immunoglobulins | Up to 24 months
  The change from baseline in IgG, IgM and IgA levels at 24 months.
Complement levels C3 and C4 | Up to 24 months
  The change from baseline in complement levels at 24 months.
Rheumatoid Factor | Up to 24 months
  The change from baseline in titer of rheumatoid factors at 24 months.
Cryoglobulins | Up to 24 months
  The change from baseline in titer of cryoglobulins at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Soledad Retamozo, MD, PhD, Principal Investigator — INICSA-Universidad Nacional de Córdoba-CONICET, Córdoba, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Retamozo S, Flores-Chavez A, Consuegra-Fernandez M, Lozano F, Ramos-Casals M, Brito-Zeron P. Cytokines as therapeutic targets in primary Sjogren syndrome. Pharmacol Ther. 2018 Apr;184:81-97. doi: 10.1016/j.pharmthera.2017.10.019. Epub 2017 Oct 29. PMID 29092775
- [Background] Kassan SS, Thomas TL, Moutsopoulos HM, Hoover R, Kimberly RP, Budman DR, Costa J, Decker JL, Chused TM. Increased risk of lymphoma in sicca syndrome. Ann Intern Med. 1978 Dec;89(6):888-92. doi: 10.7326/0003-4819-89-6-888. PMID 102228
- [Background] Jonsson R, Gordon TP, Konttinen YT. Recent advances in understanding molecular mechanisms in the pathogenesis and antibody profile of Sjogren's syndrome. Curr Rheumatol Rep. 2003 Aug;5(4):311-6. doi: 10.1007/s11926-003-0010-z. PMID 14531959
- [Background] Ioannidis JP, Vassiliou VA, Moutsopoulos HM. Long-term risk of mortality and lymphoproliferative disease and predictive classification of primary Sjogren's syndrome. Arthritis Rheum. 2002 Mar;46(3):741-7. doi: 10.1002/art.10221. PMID 11920410
- [Background] Brito-Zeron P, Retamozo S, Gheitasi H, Ramos-Casals M. Erratum to: Treating the Underlying Pathophysiology of Primary Sjogren Syndrome: Recent Advances and Future Prospects. Drugs. 2016 Dec;76(18):1799. doi: 10.1007/s40265-016-0669-x. No abstract available. PMID 27905085
- [Background] Rose T, Grutzkau A, Hirseland H, Huscher D, Dahnrich C, Dzionek A, Ozimkowski T, Schlumberger W, Enghard P, Radbruch A, Riemekasten G, Burmester GR, Hiepe F, Biesen R. IFNalpha and its response proteins, IP-10 and SIGLEC-1, are biomarkers of disease activity in systemic lupus erythematosus. Ann Rheum Dis. 2013 Oct;72(10):1639-45. doi: 10.1136/annrheumdis-2012-201586. Epub 2012 Oct 31. PMID 23117242
- [Result] Martin T, Weber JC, Levallois H, Labouret N, Soley A, Koenig S, Korganow AS, Pasquali JL. Salivary gland lymphomas in patients with Sjogren's syndrome may frequently develop from rheumatoid factor B cells. Arthritis Rheum. 2000 Apr;43(4):908-16. doi: 10.1002/1529-0131(200004)43:43.0.CO;2-K. PMID 10765938
- [Result] Quartuccio L, Baldini C, Bartoloni E, Priori R, Carubbi F, Corazza L, Alunno A, Colafrancesco S, Luciano N, Giacomelli R, Gerli R, Valesini G, Bombardieri S, De Vita S. Anti-SSA/SSB-negative Sjogren's syndrome shows a lower prevalence of lymphoproliferative manifestations, and a lower risk of lymphoma evolution. Autoimmun Rev. 2015 Nov;14(11):1019-22. doi: 10.1016/j.autrev.2015.07.002. Epub 2015 Jul 8. PMID 26162302
- [Result] Quartuccio L, Salvin S, Fabris M, Maset M, Pontarini E, Isola M, De Vita S. BLyS upregulation in Sjogren's syndrome associated with lymphoproliferative disorders, higher ESSDAI score and B-cell clonal expansion in the salivary glands. Rheumatology (Oxford). 2013 Feb;52(2):276-81. doi: 10.1093/rheumatology/kes180. Epub 2012 Aug 9. PMID 22879463
- [Result] Moore PA, Belvedere O, Orr A, Pieri K, LaFleur DW, Feng P, Soppet D, Charters M, Gentz R, Parmelee D, Li Y, Galperina O, Giri J, Roschke V, Nardelli B, Carrell J, Sosnovtseva S, Greenfield W, Ruben SM, Olsen HS, Fikes J, Hilbert DM. BLyS: member of the tumor necrosis factor family and B lymphocyte stimulator. Science. 1999 Jul 9;285(5425):260-3. doi: 10.1126/science.285.5425.260. PMID 10398604
- [Result] Schneider P, MacKay F, Steiner V, Hofmann K, Bodmer JL, Holler N, Ambrose C, Lawton P, Bixler S, Acha-Orbea H, Valmori D, Romero P, Werner-Favre C, Zubler RH, Browning JL, Tschopp J. BAFF, a novel ligand of the tumor necrosis factor family, stimulates B cell growth. J Exp Med. 1999 Jun 7;189(11):1747-56. doi: 10.1084/jem.189.11.1747. PMID 10359578
- [Result] Mariette X, Roux S, Zhang J, Bengoufa D, Lavie F, Zhou T, Kimberly R. The level of BLyS (BAFF) correlates with the titre of autoantibodies in human Sjogren's syndrome. Ann Rheum Dis. 2003 Feb;62(2):168-71. doi: 10.1136/ard.62.2.168. PMID 12525388
- [Result] Theander E, Vasaitis L, Baecklund E, Nordmark G, Warfvinge G, Liedholm R, Brokstad K, Jonsson R, Jonsson MV. Lymphoid organisation in labial salivary gland biopsies is a possible predictor for the development of malignant lymphoma in primary Sjogren's syndrome. Ann Rheum Dis. 2011 Aug;70(8):1363-8. doi: 10.1136/ard.2010.144782. PMID 21715359
- [Result] Lavie F, Miceli-Richard C, Quillard J, Roux S, Leclerc P, Mariette X. Expression of BAFF (BLyS) in T cells infiltrating labial salivary glands from patients with Sjogren's syndrome. J Pathol. 2004 Apr;202(4):496-502. doi: 10.1002/path.1533. PMID 15095277
- [Result] Szodoray P, Alex P, Jonsson MV, Knowlton N, Dozmorov I, Nakken B, Delaleu N, Jonsson R, Centola M. Distinct profiles of Sjogren's syndrome patients with ectopic salivary gland germinal centers revealed by serum cytokines and BAFF. Clin Immunol. 2005 Nov;117(2):168-76. doi: 10.1016/j.clim.2005.06.016. Epub 2005 Aug 26. PMID 16126006
- [Result] Daridon C, Devauchelle V, Hutin P, Le Berre R, Martins-Carvalho C, Bendaoud B, Dueymes M, Saraux A, Youinou P, Pers JO. Aberrant expression of BAFF by B lymphocytes infiltrating the salivary glands of patients with primary Sjogren's syndrome. Arthritis Rheum. 2007 Apr;56(4):1134-44. doi: 10.1002/art.22458. PMID 17393395
- [Result] Hjelmervik TO, Petersen K, Jonassen I, Jonsson R, Bolstad AI. Gene expression profiling of minor salivary glands clearly distinguishes primary Sjogren's syndrome patients from healthy control subjects. Arthritis Rheum. 2005 May;52(5):1534-44. doi: 10.1002/art.21006. PMID 15880807
- [Result] Wildenberg ME, van Helden-Meeuwsen CG, van de Merwe JP, Drexhage HA, Versnel MA. Systemic increase in type I interferon activity in Sjogren's syndrome: a putative role for plasmacytoid dendritic cells. Eur J Immunol. 2008 Jul;38(7):2024-33. doi: 10.1002/eji.200738008. PMID 18581327
- [Result] Brkic Z, Maria NI, van Helden-Meeuwsen CG, van de Merwe JP, van Daele PL, Dalm VA, Wildenberg ME, Beumer W, Drexhage HA, Versnel MA. Prevalence of interferon type I signature in CD14 monocytes of patients with Sjogren's syndrome and association with disease activity and BAFF gene expression. Ann Rheum Dis. 2013 May;72(5):728-35. doi: 10.1136/annrheumdis-2012-201381. Epub 2012 Jun 26. PMID 22736090
- [Result] Nezos A, Gravani F, Tassidou A, Kapsogeorgou EK, Voulgarelis M, Koutsilieris M, Crow MK, Mavragani CP. Type I and II interferon signatures in Sjogren's syndrome pathogenesis: Contributions in distinct clinical phenotypes and Sjogren's related lymphomagenesis. J Autoimmun. 2015 Sep;63:47-58. doi: 10.1016/j.jaut.2015.07.002. Epub 2015 Jul 14. PMID 26183766
- [Result] Rose T, Szelinski F, Lisney A, Reiter K, Fleischer SJ, Burmester GR, Radbruch A, Hiepe F, Grutzkau A, Biesen R, Dorner T. SIGLEC1 is a biomarker of disease activity and indicates extraglandular manifestation in primary Sjogren's syndrome. RMD Open. 2016 Dec 30;2(2):e000292. doi: 10.1136/rmdopen-2016-000292. eCollection 2016. PMID 28123773
- [Result] Barone F, Bombardieri M, Manzo A, Blades MC, Morgan PR, Challacombe SJ, Valesini G, Pitzalis C. Association of CXCL13 and CCL21 expression with the progressive organization of lymphoid-like structures in Sjogren's syndrome. Arthritis Rheum. 2005 Jun;52(6):1773-84. doi: 10.1002/art.21062. PMID 15934082